CLINICAL TRIAL: NCT06457854
Title: Real-life Experience in Brazil in Patients With Castration-resistant Prostate Cancer Treated With Olaparib+Abiraterone Observational Study Assessing Real World Clinical Endpoints and Demographic Characteristics in Patients With Castration-resistant Prostate Cancer Treated With Olaparib+Abiraterone
Brief Title: Real-life Experience in Brazil in Patients With Castration-resistant Prostate Cancer Treated With Olaparib+Abiraterone
Acronym: PROCeed-BR
Status: Withdrawn | Type: Observational
Why Stopped: 1. Decentralized sites.
  2. Lack of sites interest in the study.
  3. Super estimate of potential patient numbers.
  4. Transforming the protocol to a retrospective one could impact the study's publication timeline.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00083
Record Dates: First submitted 2024-05-23; First posted 2024-06-13 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
PROCeed is an observational study assessing real world clinical endpoints and demographic characteristics in patients with castration-resistant prostate cancer treated with Olaparib+Abiraterone.

DETAILED DESCRIPTION:
PROCeed is an observational, longitudinal study with prospective data from Brazilian participating sites, so as to generate real-world data. 10 Brazilian oncology sites are estimated to participate in the study. Each site will have participating investigators in charge and a proper technical team who will be in charge of data from each service. For this study, a convenience sample will be adopted, with an expected 2-year recruitment of 80 patients. The protocol was created in Germany and other countries could use it, with the potential for data from other countries to be pooled for analysis.

Recruitment to each subgroup will be monitored every 3 months and feasibility for continued enrolment will be assessed after 1 year of recruitment (at months 3 and 6, recruitment will be evaluated for proper site selection); if <20 patients have only been enrolled in a particular subgroup after 1 year, the study team will assess feasibility of pooling data from other countries to allow for at least 40 patients in a pooled analysis for that subgroup.

The study plans to recruit patients for no more than 2 years and to follow patients from the start of olaparib to 1 year after last patient inclusion (LPI). Data will be collected from the medical record through an electronic case report form (eCRF). Participating physicians will be responsible for ensuring that all necessary data are collected and entered in the eCRF. Data compilation will be performed by the principal investigator and statistical analysis will be performed by the statistics team appointed by the Academic Research Organization (ARO).

The target sample size of 80 patients in Brazil is based in a 24-month recruitment period. In order to avoid unnecessary imprecision for the subgroup previously exposed to a new hormonal agent, a minimum enrolment of 50% (40 patients) of the total sample size will be imposed for this subgroup. Estimation is determined based on the primary objective of the TTD event-free rate; the main measure of interest is at 6 months for patients previously exposed to NHA and 12 months for patients naïve to NHA. Assuming a 6- month TTD event-free rate is of approximately 50% for patients previously exposed to new hormonal agent, with a sample size of 40 patients in this subgroup, the precision would be +/- 15,5%.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent;
2. 18 years or older;
3. Documented histology or cytology of PCa, adenocarcinoma;
4. Documented as mCRPC;
5. Olaparib+abiraterone started after the activation of the research site.

Exclusion Criteria:

Patients participating in a clinical trial with investigational treatment for prostate cancer within 30 days before starting olaparib.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mens with documented histology or cytology of PCa and adenocarcinoma and Documented as mCRPC. This population needs to be 18 years or older. The treatment with Olaparib+abiraterone needs to start after the activation of the research site.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-02-04 (Estimated); Study Completion 2025-02-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the real-world effectiveness, measured by Time to treatment discontinuation or death, of olaparib+abiraterone in 1L Castration-resistant prostate cancer | May 2026
  Subgroup 1: patients exposed to NHA pre-olaparib+abiraterone initiation; Subgroup 2: patients not exposed to NHA pre-olaparib+abiraterone initiation. The main measure of interest is Time to treatment discontinuation or death (TTD) with corresponding 95% confidence intervals in 6-month and 12-month timepoints for subgroup 1 and subgroup 2, respectively. This analysis will be performed only in patients with Castration-resistant prostate cancer(mCRPC) 1L. Patients exposed to abiraterone pre- olaparib+abiraterone initiation will be excluded from this primary analysis

SECONDARY OUTCOMES:
Describe the demographic and clinical characteristics of Castration-resistant prostate cancer patients treated with olaparib+abiraterone in the general population and also in each population. | May 2026
  Subgroup 1: patients exposed to NHA pre-olaparib+abiraterone initiation; Subgroup 2: patients not exposed to NHA pre-olaparib+abiraterone initiation. This analysis will be performed in Castration-resistant prostate cancer (mCRPC) 1L patients (base case analysis) and in all patients with mCRPC (sensitivity analysis).
Describe the treatments received before and after olaparib+abiraterone in general population and also in each population. | May 2026
  Subgroup 1: patients exposed to NHA pre-olaparib+abiraterone initiation; Subgroup 2: patients not exposed to NHA pre-olaparib+abiraterone initiation. This analysis will be performed in mCRPC 1L patients (base case analysis) and in all patients with mCRPC (sensitivity analysis).
To evaluate Time to first subsequent therapy or death in patients with Castration-resistant prostate cancer treated with olaparib+abiraterone in general population and also in each population. | May 2026
  Subgroup 1: patients exposed to NHA pre-olaparib+abiraterone initiation; Subgroup 2: patients not exposed to NHA pre-olaparib+abiraterone initiation. This analysis will be performed in mCRPC 1L patients (base case analysis) and in all patients with mCRPC (sensitivity analysis).
To describe the demographic data, clinical characteristics, previous and subsequent treatments of patients with mCRPC treated with olaparib+abiraterone in overall cohort and in subgroups 1 and 2, additionally stratified by BRCA/HRR mutation status. | May 2026
  This analysis will be performed in mCRPC 1L patients (base case analysis) and in all patients with mCRPC (sensitivity analysis).

OTHER OUTCOMES:
To evaluate the real world effectiveness, measured by Time to treatment discontinuation or death, of olaparib+abiraterone in 1L mCRPC | May 2026
  Subgroup 1: patients exposed to NHA pre-olaparib+abiraterone initiation (TTD rate (event- free) with corresponding 95% confidence intervals in 3, 9, 12 and 24-month timepoints and median TTD); Subgroup 2: patients not exposed to NHA pre-olaparib+abiraterone initiation. (TTD rate (event-free) with corresponding 95% confidence intervals in 3, 6, 9 and 24 -month timepoints and median TTD). Patients exposed to abiraterone pre-olaparib+abiraterone initiation will be excluded from this exploratory objective analysis. This analysis will also be performed only in patients with 1L mCRPC.
To evaluate additional clinical outcomes (OS, rwPFS) in general population and also in each population | May 2026
  Subgroup 1: patients exposed to NHA pre-olaparib+abiraterone initiation; Subgroup 2: patients not exposed to pre-olaparib+abiraterone initiation. Patients exposed to abiraterone pre-olaparib+abiraterone initiation will be excluded from this analysis. This analysis will also be performed only in patients with 1L mCRPC.
Describe the dosage in patients treated with the combination of olaparib+abiraterone in general population and also in each population | May 2026
  Subgroup 1: patients exposed to NHA pre-olaparib+abiraterone initiation; Subgroup 2: patients not exposed to NHA pre-olaparib+abiraterone initiation. This analysis will be performed in mCRPC 1L patients (base case analysis) and in all patients with mCRPC (sensitivity analysis).
Describe the reasons for dose change/discontinuation in patients treated with the combination of Olaparib+Abiraterone in general population and also in each population | May 2026
  Subgroup 1: patients exposed to NHA pre-olaparib+abiraterone initiation; Subgroup 2: patients not exposed to NHA pre-olaparib+abiraterone initiation. This analysis will be performed in mCRPC 1L patients (base case analysis) and in all patients with mCRPC (sensitivity analysis).
To evaluate the PSA25 and PSA50 response with an evaluation tool to predict the practical clinical activity in the real world. | May 2026
  This analysis will be performed only in patients with mCRPC 1L.
To evaluate the time to progression of PSA. | May 2026
  This analysis will be performed only in patients with mCRPC 1L.

CONTACTS AND LOCATIONS:
Overall Officials: Henrique Helber, Study Chair — Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein Centro de Ensino e Pesquisa Albert Einstein
Locations (5):
- Brazil (5):
  - Clínica AMO, Salvador, Estado de Bahia
  - Liga Norte Rio Grandense Contra o Câncer, Natal, Rio Grande do Norte
  - Clínica Viver, Santa Maria, Rio Grande do Sul
  - Hospital Alemão Oswaldo Cruz, São Paulo
  - Hospital Albert Einstein, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/